CLINICAL TRIAL: NCT02801370
Title: A Prospective, Randomized, Double-Blind, Sham-Controlled, Multicenter, Phase 3 Study of OTO-201 Given as a Single Administration for Treatment of Acute Otitis Externa
Brief Title: Phase 3 Study of OTO-201 in Acute Otitis Externa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 201-201609
Record Dates: First submitted 2016-06-13; First posted 2016-06-15 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Acute Otitis Externa; Swimmer's Ear
MeSH Terms: conditions — Otitis Externa | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OTO-201 (Experimental)
  Interventions: Drug: 12 mg ciprofloxacin
- Control (Sham Comparator)
  Interventions: Drug: Sham Control

INTERVENTIONS:
Drug: 12 mg ciprofloxacin — Single administration of OTO-201
  Other Names: OTIPRIO
  Arms: OTO-201
Drug: Sham Control — Simulated, single adminstration
  Arms: Control

SUMMARY:
This is a prospective, randomized, double-blind, sham-controlled, multicenter, Phase 3 study in which eligible subjects with acute otitis externa (AOE) will be randomized to receive a single administration of either 12 mg OTO-201 or Sham-Control (empty syringe) to the external auditory canal of the affected ear(s).

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject is a male or female age 6 months or older
* Subject has a clinical diagnosis of unilateral or bilateral acute otitis externa
* Subject or subject's caregiver is willing to comply with the protocol and attend all study visits

Exclusion Criteria includes, but is not limited to:

* Subject has tympanic membrane perforation
* Subject has eczematoid otitis externa
* Subject has diabetes mellitus

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Chair — Otonomy, Inc.
Locations (2):
- Call Otonomy call center for trial locations, San Diego, California, United States
- Call Otonomy call center for trial locations, Saskatoon, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 12 mg OTO-201: 12 mg ciprofloxacin: single administration
Period: Overall Study
Arm/Group | 12 mg OTO-201 | Control
Started | 130 | 132
Completed | 123 | 132
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Population: 262 subjects randomized (132 sham, 130 OTO-201). 2 sham subjects positive for Group A strep and not in ITT population (Baseline characteristics and efficacy) leaving 130 sham, 130 OTO-201. ITT subjects analyzed as randomized. Safety population (AE/SAE) analyzed by what was received (132 sham, 127 OTO-201) regardless of culture, but had be dosed.
Groups:
- Control: Sham Control: Simulated, single administration
- Total: Total of all reporting groups
Arm/Group | 12 mg OTO-201 | Control | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.724 (20.5866) | 34.796 (19.2708) | 35.760 (19.9244)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 55 | 55 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 43 | 84
  Not Hispanic or Latino | 87 | 86 | 173
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 14 | 15 | 29
  White | 111 | 109 | 220
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 130 | 130 | 260

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Considered a Clinical Cure at Day 8
Description: Clinical Signs (edema, erythema, otorrhea and otalgia) all had a score of 0 at Day 15. Each sign was graded as follows:
  None = 0 Mild = 1 Moderate = 2 Severe = 3
Time Frame: At Day 8 (1 week after dosing)
Population: Intent-to-treat analysis set: All subjects who were randomized and did not have Group A Streptococci cultured on Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | 12 mg OTO-201 | Control
Number analyzed (Participants) | 130 | 130
Participants | 91 | 63

2. Secondary Outcome: Number of Subjects Considered a Clinical Cure at Day 15
Description: as for outcome 1
Time Frame: At Day 15 (2 weeks after dosing)
Population: Intent-to-treat analysis set: All subjects who were randomized and and did not have Group A Streptococci cultured on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 mg OTO-201 | Control
Number analyzed (Participants) | 130 | 130
Participants | 97 | 69

ADVERSE EVENTS:
Time Frame: Adverse events were reported during dosing and up to 1 month following dosing.
Arm/Group | 12 mg OTO-201 | Control
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/132
Other Adverse Events (participants affected / at risk) | 12/127 | 18/132
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12 mg OTO-201 (N=127) | Control (N=132)
Otitis externa (Infections and infestations) | 3 | 9
Ear Pain (Ear and labyrinth disorders) | 3 | 3
Ear pruritis (Ear and labyrinth disorders) | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication subject to Sponsor consent.